CLINICAL TRIAL: NCT05382871
Title: A Randomized, Double-Blinded, Cohort Clinical Study on Evaluating the Safety and Immunogenicity of Sequential Immunization of Two Doses of BIBP Inactivated COVID-19 Vaccine (Omicron), WIBP Inactivated COVID-19 Vaccine (Omicron) or Inactivated COVID-19 Vaccine (Prototype) in Population Aged 18 Years and Above Who Have Completed Two or Three Doses of Inactivated or mRNA Vaccine
Brief Title: Sequential Immunization of Two Doses of Inactivated COVID-19 Vaccine (Omicron) in Vaccinated Population Aged 18 Years and Above
Acronym: COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Wuhan Institute of Biological Products Co., Ltd (Industry); The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CNBG-O-2022002
Record Dates: First submitted 2022-05-17; First posted 2022-05-19 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1: BIBP Inactivated COVID-19 vaccine (Omicron) (Experimental): subjects will be blinded and receive two doses of BIBP Inactivated COVID-19 vaccine (Omicron) with 28 days apart more than 3 months after 2 or 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: BIBP Omicron Inactivated COVID-19 vaccine (Vero Cell)
- 2: WIBP Inactivated COVID-19 vaccine (Omicron) (Experimental): subjects will be blinded and receive two doses of WIBP Inactivated COVID-19 vaccine (Omicron) with 28 days apart more than 3 months after 2 or 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: WIBP Omicron Inactivated COVID-19 vaccine (Vero Cell)
- 3：BIBP Inactivated COVID-19 vaccine (Omicron) (Experimental): subjects will be blinded and receive two doses of BIBP Inactivated COVID-19 vaccine (Omicron) with 28 days apart more than 3 months after 2 or 3 doses of COVID-19 mRNA vaccine
  Interventions: Biological: BIBP Omicron Inactivated COVID-19 vaccine (Vero Cell)
- 4: WIBP Inactivated COVID-19 vaccine (Omicron) (Experimental): subjects will be blinded and receive two doses of WIBP Inactivated COVID-19 vaccine (Omicron) with 28 days apart more than 3 months after 2 or 3 doses of COVID-19 mRNA vaccine
  Interventions: Biological: WIBP Omicron Inactivated COVID-19 vaccine (Vero Cell)
- 5：Inactivated COVID-19 Vaccine (prototype) (Active Comparator): subjects will be blinded and receive two doses of Inactivated COVID-19 Vaccine (prototype) with 28 days apart more than 3 months after 2 or 3 doses of inactivated COVID-19 vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- 6：Inactivated COVID-19 Vaccine (prototype) (Active Comparator): subjects will be blinded and receive two doses of Inactivated COVID-19 Vaccine (prototype) with 28 days apart more than 3 months after 2 or 3 doses of COVID-19 mRNA vaccine
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: BIBP Omicron Inactivated COVID-19 vaccine (Vero Cell) — intramuscular injection in the deltoid muscle
  Arms: 1: BIBP Inactivated COVID-19 vaccine (Omicron); 3：BIBP Inactivated COVID-19 vaccine (Omicron)
Biological: WIBP Omicron Inactivated COVID-19 vaccine (Vero Cell) — intramuscular injection in the deltoid muscle
  Arms: 2: WIBP Inactivated COVID-19 vaccine (Omicron); 4: WIBP Inactivated COVID-19 vaccine (Omicron)
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — intramuscular injection in the deltoid muscle
  Arms: 5：Inactivated COVID-19 Vaccine (prototype); 6：Inactivated COVID-19 Vaccine (prototype)

SUMMARY:
This trial adopts a randomized, double-blind and positive control design, it is planned to recruit 1800 healthy participants who have been vaccinated with 2/3 doses of COVID-19 inactivated vaccine or mRNA vaccine for 3 months. The participants will be divided into two strata according to the types of vaccines administered, including 900 participants of COVID-19 inactivated vaccine and 900 participants of mRNA vaccine. According to the ratio of 1:1:1, each stratum was randomly assigned to three groups: sequential BIBP- COVID-19 inactivated vaccine (Omicron), WIBP-COVID-19 inactivated vaccine (Omicron) or COVID-19 inactivated vaccine (prototype strain). And according to D0, D28 immunization schedule, two doses of corresponding group vaccines are sequentially administered.

ELIGIBILITY:
Inclusion Criteria:

* Age range: populations aged 18 years and above.
* Judged by the investigator that the health condition is well after inquiry and physical examination.
* Vaccinated with 2 doses/3 doses of inactivated COVID-19 vaccine or mRNA vaccine for ≥ 3 months.
* Female participants who are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 7 months after enrollment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* During the whole follow-up period of the study, be able and willing to complete the whole prescribed study plan.
* With self ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and is able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Confirmed cases, suspected cases or asymptomatic cases of COVID-19;
* With a history of Severe Acute Respiratory Syndrome (SARS) and Middle East Respiratory Syndrome (MERS) (self-report, on-site inquiry);
* Has vaccinated with one or four doses and above COVID-19 vaccine;
* Axillary temperature ≥37.3℃ (Tympanic temperature ≥ 37.6 ℃);
* Previous allergic reactions to drug or vaccination (such as acute allergic reactions, urticaria, eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to known components of COVID-19 vaccine (self-report, onsite enquiry);
* Have a history of hospital-diagnosed thrombocytopenia or other coagulation disorders (self-report, onsite enquiry);
* With known immunological impairment or immunocompromised diagnosed by the hospital (self-report, onsite enquiry);
* Have an uncontrolled epilepsy and other progressive neurological diseases or a history of Guillain-Barre syndrome (self-report, onsite enquiry);
* Received whole blood, plasma and immunoglobulin therapy within 1 month (self-report, onsite enquiry);
* Known or suspected severe illness includes: respiratory illness, acute infection or active attacks of chronic illness, liver and kidney disease, severe diabetes mellitus, malignant tumor, infectious or allergic skin disease, Human Immunodeficiency Virus (HIV) infection (self-report, onsite enquiry, provide test report if available);
* With hospital-diagnosed serious cardiovascular diseases (cardiopulmonary failure, drug-uncontrolled hypertension (physical examination of systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg), acute attacks of chronic respiratory illness (self-report, onsite enquiry);
* Received live attenuated vaccines within 1 month before vaccination (self-report, onsite enquiry);
* Received inactivated vaccines within 14 days before vaccination (self-report, onsite enquiry);
* Participating or planning to participate in other interventional vaccine clinical trials during this study
* Other vaccination-related contraindications considered by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1804 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-07-27 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The Geometric Mean Titer （GMT） of anti-omicron neutralizing antibody | 28 days after sequential vaccination of 2 doses
The 4-fold rise rate of anti-omicron neutralizing antibody | 28 days after sequential vaccination of 2 doses

SECONDARY OUTCOMES:
The GMT of anti-omicron neutralizing antibody | 14 days after sequential vaccination of 2 doses
The 4-fold rise rate of anti-omicron neutralizing antibody | 14 days after sequential vaccination of 2 doses
Specific cellular immune response | within 28 days after vaccination
The GMT of anti-omicron Immunoglobulin G (IgG) antibody | 28 days after sequential vaccination of 2 doses
The proportions of neutralizing antibody titer ≥ 1: 16, ≥ 1: 32 and ≥ 1: 64 | 28 days after sequential vaccination of 2 doses
The proportion of subjects with neutralizing antibody GMT ≥1:16，≥1:32 and ≥1:64 | on 3rd month, 6th month, 9th month, and 12th month after vaccination
The incidence of any adverse reactions/events | 28 days after each immunization
The incidence of serious adverse events (SAE) and adverse events special interest (AESI) | from 1st booster dose and up to 6 months following 2nd booster dose

OTHER OUTCOMES:
The incidence of COVID-19 cases , including severe cases and deaths accompanied by COVID-19 | From 14 day after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Hung, Clinical Professor, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No